CLINICAL TRIAL: NCT04355832
Title: Reducing Hypoglycemic, Pro-coagulant and Pro-atherothrombotic Responses and Preventing Hypoglycemia Associated Autonomic Failure in Type 1 DM. The Effects of Glucagon-like Peptide-1
Brief Title: Glucagon-like Peptide-1 in Type 1 Diabetes
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: We were unable to obtain GLP-1
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Stephen N. Davis, MBBS, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HP-00090856
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Type1 Diabetes Mellitus
MeSH Terms: interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo 1 (Placebo Comparator): The participants will be randomized to placebo infusion.
  Interventions: Drug: Placebos
- Placebo 2 (Placebo Comparator): The participants will be randomized to placebo infusion.
  Interventions: Drug: Placebos
- GLP-1 (Experimental): The participants will be randomized to Glucagon-like peptide-1 infusion.
  Interventions: Drug: Glucagon-like peptide-1

INTERVENTIONS:
Drug: Glucagon-like peptide-1 — Infusion of Glucagon-like peptide-1
  Arms: GLP-1
Drug: Placebos — Infusion of normal saline solution that will mimic Glucagon-like peptide-1
  Arms: Placebo 1; Placebo 2

SUMMARY:
The hypotheses to be tested in this application is: GLP-1 will acutely protect arterial endothelial function and reduce pro-atherothrombotic and pro-coagulant effects of repeated hypoglycemia in T1DM.

DETAILED DESCRIPTION:
The naturally occurring hormone GLP-1 when co-administered during hypoglycemia (low blood sugar) in non-diabetic individuals can reduce the deleterious effects of hypoglycemia on the vasculature. We have shown that IV infusion of GLP-1 during a single moderate episode of hypoglycemia can preserve endothelial function and protect the vasculature from pro-coagulant and pro-inflammatory effects in healthy individuals.

It is unknown whether GLP-1 could protect the vasculature during episodes of repeated hypoglycemia and whether GLP-1 would have protective effects in T1DM individuals.

ELIGIBILITY:
Inclusion Criteria:

* 40 (20 males, 20 females) individuals with type 1 diabetes aged 18-50 yr.
* HbA1c < 11.0%
* Body mass index < 40kg • m-2
* No clinically diagnosed diabetic tissue complications (i.e. history of retinopathy, neuropathy, stasis ulcers, etc)

Exclusion Criteria:

* Subjects unable to give voluntary informed consent
* Pregnancy
* Subjects on anticoagulant drugs, anemic or with known bleeding diatheses
* Subjects taking any of the following medications will be excluded: non-selective beta blockers,
* sedative-hypnotics, anticonvulsants, antiparkinsonian drugs, antipsychotics, antidepressants,
* mood stabilizers, CNS stimulants, opioids, hallucinogens
* Subjects unwillingness or inability to comply with approved contraception measures
* Subjects with a history of severe uncontrolled hypertension (i.e., blood pressure greater than 160/100), heart disease, cerebrovascular incidents
* Clinically significant cardiac abnormalities (e.g. heart failure, arrhythmias, ischemic tachycardia, S-T segment deviations, etc.) from history or from cardiac stress testing in subjects ≥ 40 years old.
* Pneumonia
* Hepatic failure /jaundice
* Abnormal results following screening tests and physical examination that are clinically significant
* Acute cerebrovascular/ neurological deficit
* Fever greater than 38.0 C
* Screening Laboratory Tests Exclusion Criteria
* Hematocrit lower than 32
* WBC lower than 3 thou/ul or greater than 14 thou/ul
* Liver function tests: SGOT and SGPT greater than twice upper limit of normal range (i.e. > 80 U/L)
* TBil > 2 mg/dl
* Creatinine > 1.6 mg/dl
* Alkaline phosphatase > 150U/L
* Hepatic transaminase > 2x normal

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Change in the level of catecholamines in plasma | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No